# NON INTERVENTIONAL STUDY STATISTICAL ANALYSIS REPORT (POST-MARKET CLINICAL FOLLOW-UP STUDY)

### **SPONSOR**

Pierre Fabre Médicament Les Cauquillous 815000 LAVAUR, France

### Toux Petit (C1735)

The Performance and Safety of Petit Drill in the French Paediatric Population: a post-market clinical follow-up study

### **Biostatistician**

Romain SCHUELLER CEN (CRO) 18, rue Pauline Kergomard 21000 DIJON, France

Data-management Nhu-Anh TRAN CEN (CRO)

Medical writing Christine JUHEL CEN (CRO)

Date: May 14, 2025 CEN Version: v1.0 PF Version: Final Version

C1735\_RAS\_1.0\_RNSR\_20250514.docx

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>2</b> on <b>81</b> |
|---|---|---|---|
|---|---|---|---|

### **HISTORY OF VERSIONS**

| N°<br>Pierre<br>Fabre | N° CEN | Date | Reasons for changes |
|---|---|---|---|
| Draft 1 | v0.1 | 01/04/2025 | Creation of the document: RNSR |
| Draft 1 | v0.2 | 30/04/2025 | New version sent to CEN by Kalaivani RUHIER |
| Draft 1 | v0.3 | 05/05/2025 | New version CEN RNSR (after incorporating the changes requested by KIRR) |
| Draft 1 | v0.4 | 13/05/2025 | New version sent to CEN by Kalaivani RUHIER |
| Draft 1 | v0.5 | 13/05/2025 | New version CEN RNSR (after incorporating the changes requested by KIRR) with track changes |
| Draft 1 | v0.6 | 13/05/2025 | New version sent to CEN by Kalaivani RUHIER |
| Final<br>Version | V1.0 | 13/05/2025 | Final version CEN RNSR (after incorporating last changes requested by KIRR) |

### APPROVAL OF THE STATISTICAL ANALYSIS REPORT

| PROTOCOL TITLE | The Performance and Safety of Petit Drill in the French Paediatric Population: a post-market clinical follow-up. |
|---|---|
| VERSION OF PROTOCOL | Final version v6.0 – 2024/03/26 |
| VERSION OF THE STATISTICAL ANALYSIS PLAN | Final version v1.0 – 2025/03/31 |

STATISTICAL ANALYSIS REPORT

Final version - 2025/05/14

| FUNCTION | NAME,<br>OFFICE | RESPONSABILITY | SIGNATURE/DATE |
|---|---|---|---|
| Project Load | Cécile<br>HAUVILLE | | Signé par : Cuile HAUVILLE |
| Project Lead | Pierre Fabre<br>Médicament | Approver | Nom du signataire : Cécile HAUVILLE Motif de la signature : J'approuve ce document Heure de signature : 14-mai-2025 09:49 CEST 426B097E7AD340AAAB9D1AB5092D99ED |
| Medical<br>Advisor | Didier<br>JUNQUERO | Approver | Signé par: Didier Junquero |
| global | Pierre Fabre<br>Médicament | Approver | Nom du signataire : Didier Junquero Motif de la signature : J'approuve ce document Heure de signature : 14-mai-2025 09:54 CEST 280A37180FBB41F99513AFC7AFAC41B3 |
| Biostatistician | Kalaivani<br>RUHIER | Approver | Signé par :<br>kalaivani KUHEK |
| IVIDATA | Pierre Fabre<br>Médicament | | Nom du signataire : Kalaivani RUHIER Motif de la signature : J'approuve ce document Heure de signature : 14-mai-2025 11:39 CEST C5CA9E9FE9A648C185DE5F5CF68FF134 |
| Medical | Christine<br>JUHEL | Author | Signé par : (Unistine JUHE) |
| writing | CEN | | Nom du signataire : Christine JUHEL Motif de la signature : J'ai examiné ce document Heure de signature : 14-mai-2025 12:14 CEST 4430C79AA9884546807FD2A8FE73CA06 |
| Riostatistician | Romain<br>SCHUELLER | Author | Signé par : Romain SCHUEUER |
| Biostatistician | CEN | Autioi | Nom du signataire : Romain SCHUELLER Motif de la signature : J'ai rédigé ce document Heure de signature : 14-mai-2025 09:49 CEST 8047B0B45A8442B49337D548390FDAB2 |

### **SOMMAIRE**

| Н | ISTOR | RY OF VERSIONS | 2 |
|---|---|---|---|
| Α | PPRO | VAL OF THE STATISTICAL ANALYSIS REPORT | 3 |
| S | OMMA | AIRE | 4 |
| 1 | ABI | BREVIATION | 6 |
| 2 | | RODUCTION | |
| _ | 2.1 | Study objectives | |
| | 2.1.1 | | <b>ອ</b> |
| | 2.1. | | |
| | 2.1.3 | , , | |
| | | Study methods | |
| | 2.2.1 | • | |
| | 2.2.2 | | |
| | | 2.2.1 Inclusion criteria | |
| | | 2.2.2 Exclusion criteria | |
| | 2.2.3 | | |
| | 2.2.4 | | .11 |
| | 2.2.5 | | |
| | | Statistical methodology | |
| 3 | IND | EX | 15 |
| | 3.1 | Summary Tables index | .15 |
| | 3.2 | Tables index | |
| | 3.3 | Figures index | |
| | 3.4 | Listings index | |
| 4 | DEG | SULTS | 17 |
| 4 | | | |
| | 4.1<br>4.2 | Description of Study Conduct | |
| | 4.2 | Children not pre-selected by pharmacists (Register 1) and not included by investigator (Register 2) | |
| | 4.3 | Disposition of patients | |
| | 4.3 | Clinical and sociodemographic characteristics of children using Petit D | |
| | 4.4 | (FAS population) | |
| | 4.4.1 | · · · · · · | |
| | 4.4.2 | | |
| | 4.4.3 | | |
| | 4.4.4 | · | |
| | 4.4.5 | | |
| | 7.7.0 | population) | |
| | 4.5 | Concomitant treatments during follow up (FAS population) | .39 |
| | 4.6 | Primary endpoint - Change in PCQ total score (PERFORMANCE POPULATION | ON) |
| | | | .40 |
| | 4.7 | Secondary outcome - PCQ items (PERFORMANCE POPULATION) | |
| | 4.8 | Secondary outcome - Daily cough severity (VAS) (PERFORMAN | |
| | | POPULATION*) | .54 |
| | 4.9 | Secondary outcome - Change in PAC-QoL total score* | .57 |
| | 4.10 | Secondary outcome - PAC-QoL items* | |
| | 4.11 | Secondary outcome - Adherence (FAS population) | |
| | 4.12 | Secondary outcome - Satisfaction questionnaire (FAS population) | |
| | 4.13 | Secondary outcome: Safety evaluation - SAFETY population | .76 |

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>5</b> on <b>81</b> |
|---|---|---|---|
| 4.14 Se | condary outcome: Device deficie | encies (SAFFTY) | 8 |
| 7.17 | condary outcome. Device denote | indices (OAI ETT) | |

| C1735 Statistical Analysis Report | 14/05/2025 | Page <b>6</b> on <b>81</b> |
|-----------------------------------|------------|----------------------------|
|-----------------------------------|------------|----------------------------|

### 1 ABBREVIATION

| ADE | Adverse Device Effect |
|---|---|
| AE | Adverse Event |
| ANSM | Agence Nationale de sécurité du médicament et des produits de santé |
| ВМІ | Body Mass Index |
| CI | Confidence Interval |
| CIR | Clinical Investigation Report |
| CIP | Clinical Investigation Plan |
| CPP | Comité de Protection des Personnes |
| CRO | Clinical Research Organization |
| CSS | Cough Symptom Score |
| D0 | The day before treatment initiation |
| D1 | The first day of treatment initiation |
| D2 | The second day of treatment initiation |
| D3 | Third day of treatment |
| DD | Device Deficiencies |
| EC | Ethics Committee |
| eCRF | Electronic Case Report Form |
| FAS | Full Analysis Set |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GDPR | General Data Protection Regulation |
| ICF | Informed Consent Form |
| IFU | Instructions for Use |
| MCID | Minimum Clinically Important Difference |
| MD | Medical Device |
| MDCG | Medical Device Coordination Group guidelines |
| MDR | Medical Device Regulation |
| MHRA | Medicines and Healthcare products Regulatory Agency |
| OTC | Over-the-Counter |
| PAC-QoL | Parent-proxy Children's Acute Cough-specific QoL Questionnaire |
| PCQ | Pediatric Cough Questionnaire |
| PI | Principal investigator of the site |
| PMCF | Post-Market Clinical Follow-up |
| PRO | Patient Reported Outcome |
| QoL | Quality of Life |
| QC | Quality Control |
| SAE | Serious Adverse Event |

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>7</b> on <b>81</b> |
|---|---|---|---|
| SADE Serious Adverse Device Effect | | | |
| SAP | Statistical Analysis Plan | | |
| SD | Standard Deviation | | |
| URTI | Upper Respiratory Tract Infection | | |
| VAS | Visual Analogue Scale | | |
| WHO | World Health Organisation | | |

| C1735 Statistical Analysis Report | 14/05/2025 | Page <b>8</b> on <b>81</b> |
|-----------------------------------|------------|----------------------------|
|-----------------------------------|------------|----------------------------|

### 2 INTRODUCTION

This present document refers to the final statistical analysis report of the Touxpetit study Its objective is to present the results of all the pre-specified study objectives. This report has been produced in accordance with all the approved documents prior to the database lock, including:

- Synopsis Version 6.0, dated 06/02/2024.
- Protocol Version 6.0, dated 26/03/2024.
- Annotated CRF Version 3.0, one annotated eCRF for data collected in the Nurstrial application dated on 19/03/202 and one annotated eCRF for data collected in the ENNOV eCRF on 08/03/2024.
- Statistical Analysis Plan (SAP, v1.0 dated 31/03/2025).
- Data review report (DR, v1.0 dated 31/03/2025).

The data was reviewed on March 12<sup>th</sup>, 2025, and the database lock was performed in March 31<sup>st</sup>, 2025. The results presented in this document are reported in the following formats: tables, figures, and listings, all produced from the derived database. The TFLs were generated and edited using SAS version 9.4.

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>9</b> on <b>81</b> |
|---|---|---|---|
|---|---|---|---|

### 2.1 Study objectives

### 2.1.1 Primary objective

To assess the performance of the Petit Drill medical device in the treatment of throat irritation (sore throat) associated with dry cough in infants starting at 6 months of age and in children up to 6 years of age.

### 2.1.2 Secondary objectives

• SO1. To describe the clinical and sociodemographic characteristics of children using Petit Drill.

The following secondary objectives described the performance and clinical benefit of Petit Drill in terms of:

- SO2. Changes in nightly cough frequency, severity, bothersome for the child, and ability to sleep for child and parent(s) throughout the 3 day-treatment;
- SO3. Changes in daily cough severity;
- SO4. Evolution of Quality of life.

The following secondary objectives will describe the use and safety of Petit Drill:

- SO5. Adherence to use of Petit Drill Syrup;
- SO6. Parents' satisfaction with Petit Drill use;
- SO7. Safety of the Petit Drill medical device in infants aged from 6 months to children up to 6 years of age.

### 2.1.3 Exploratory objectives

- SO8. To describe the dispensing modalities of Petit Drill by age group;
- SO9. To describe the study objectives (except SO8) according to child's range of age.

| C1735 Statistical Analysis Report | 14/05/2025 | Page <b>10</b> on <b>81</b> |
|-----------------------------------|------------|-----------------------------|
| C1735 Statistical Analysis Report | 14/05/2025 | Page 10 on 61 |

### 2.2 Study methods

### 2.2.1 Study design

This is an observational, prospective French national, monocentric, single-arm, descriptive clinical investigation with pre-screened patients, for whom we have not to mandate or recommend any additional interventions or in-person visits. Patients continued to be treated as per routine practice.

### 2.2.2 Inclusion/exclusion criteria

The entry criteria have been chosen in such a way as to allow selection of the population targeted by Petit Drill when used for its intended purpose. These criteria also had to ensure that the study could be carried out effectively and that the regulations were complied with. Finally, most of exclusion criteria were supposed to limit confounding factor.

Criteria hereafter were necessary and sufficient to meet the objectives of this study.

### 2.2.2.1 Inclusion criteria

Children meeting the following inclusion criteria were included:

- IC1. Boys or girls, 6 months to 6 years of age;
- IC2. With one of his/her parents/legal guardian purchases Petit Drill in a participating pharmacy in accordance with recommendations for use (regarding age and type of cough);
- IC3. For infants between 6 months and 12 months of age a confirmed prescription from a treating physician;
- IC4. With an acute cough lasting less than 48 hours
- IC5. With a score ≥ 3 at least for 3 of the 5 items of PCQ, (based on assessment of the night before inclusion);
- IC6. For whom child-minding will allow to respect the recommended daily doses\* of Petit Drill during the 3 day-treatment;
- IC7. With a parent/legal guardian having a smartphone allowing using the ePRO App. NursTrial<sup>®</sup>;
- IC8. With a parent/legal guardian able to understand and to complete to the questionnaires in timely manner;
- IC9. With parent(s)/legal guardian who provide their signed informed consent for the child's enrolment in the study.

<sup>\* 2-4</sup> doses on D1, then 3 to 4 doses on D2 and D3, including one of the daily doses taken at bedtime.

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>11</b> on <b>81</b> |
|---|---|---|---|

### 2.2.2.2 Exclusion criteria

Children meeting one of the following exclusion criteria were excluded:

- EC1. Presenting with one of the following conditions:
  - Chronic respiratory illness such as asthma, recurrent wheezing associated to viral infections and bronchitis;
  - Lower respiratory infections, such as bronchitis, bronchiolitis, and pneumonia;
  - o Tonsillitis, otitis, or sinusitis;
  - Persistent cough lasting more than 3 weeks, whatever the etiology;
  - o Gastrointestinal pathology, involving vomiting, nausea, or diarrhoea.
- EC2. With ongoing use of paracetamol, and/or homeopathic products against cough;
- EC3. Having had corticosteroid treatment, antibiotics, antihistaminic or any cough medication (such as, but not limited to, Phytoxil, Arkotoux) in the previous 15 days since inclusion;
- EC4. With a brother/sister already included in the present clinical investigation\*;
- EC5. Enrolled in another clinical trial or being in a period of exclusion from a previous clinical trial.

### 2.2.3 Study populations

**Pre-screen-failed/refusal register 1 (Pharmacist register)**: pre-screening log completed by the pharmacist for children not taking part in the study with the collection of the following data: age, sex and reason for non-inclusion to the investigation.

**Screen-failed register 2 (Investigator register)**: pre-screening log will be completed by the investigator for children not taking part in the study including the following data: age, sex, reason for non-inclusion in the investigation, date of dry cough onset and the PCQ-score (based on the recall of the night prior inclusion).

**Full Analysis Set (FAS) population\***: The analysis population will consist of patients who have been included in this clinical investigation after fulfilling all eligibility criteria.

**Safety population**: The safety population will include all patients from the FAS population who have used Petit Drill at least once.

**Performance population**\*: The performance population will consist of all patients from the safety population without any major deviation from the protocol\*\* and for whom at least one evaluation of the primary outcome is available after treatment initiation (baseline and the last assessment) and whose parent(s) or legal guardian did not withdraw their consent at any time.

### Note:

\*FAS population refers to the analysis population and performance population refers to the evaluable population.

\*\*Taking treatments prohibited by the protocol before and during the study was considered a major deviation.

### 2.2.4 Study subpopulations

2 subpopulations based on age were defined as follow:

- Patients aged from 6 months to 12 months old (12 included): [6 months -12 months];
- Patients aged from 12 (12 not included) months old to 6 years old: ]12months 6 years].

These two subpopulations will only be used to meet the exploratory objective SO8 of the protocol.

<sup>\*</sup> If several children were eligible in the same household, only one may was enrolled at random.

| C1735 Statistical Analysis Report | 14/05/2025 | Page <b>12</b> on <b>81</b> |
|-----------------------------------|------------|-----------------------------|
|-----------------------------------|------------|-----------------------------|

### 2.2.5 Subgroup definition

Age subgroup was defined as follow:

- Patients aged from 6 months to 24 months old (24 not included): [6 months 24 months[;
- Patients aged from 24 months (24 included) old to 6 years old: [24 months 6 years].

All the objectives except the exploratory objective SO8 were reproduced by age subgroup.

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>13</b> on <b>81</b> |
|---|---|---|---|

# 2.3 Statistical methodology

The statistical analysis to be conducted following the premature termination of the study, along with the derivation rules, are fully detailed in the final version of SAP dated on March 31st, 2025. The final analysis is exclusively descriptive.

The table below provides a summary of the analyses that were performed for the final analysis following the study's early termination.

Summary\_Table 1: Analyses performed after premature study termination

| 0.0000000000000000000000000000000000000 | | | | | |
|---|---|---|---|---|---|
| Analyses performed | Scheduled TFLs (before the premature study termination) | Based on<br>planned<br>TFLs (1) or<br>new TFLs<br>(2) | Type of TFLs to be produced | TFLs performed (after the premature study termination) | Population concerned |
| Description of Study conduct (key dates/durations) | Scheduled_Table 1 | 1 | Table | Table 1 | Full analysis population |
| Children not pre-selected by pharmacists (Register 1) and not included by the investigator (Register 2) | Scheduled_Table 2 and Scheduled_Table 3 | 1 & 2 | Table | Table 2 and Listing 1, Table 3 and listing 2 | Full analysis<br>population |
| Disposition of patients - Overall population | Scheduled_Table 4_and<br>Scheduled_Figure 1 | 1 | Table & Figure | Table 4 and Figure 1 | Full analysis population |
| Disposition of patients - Subgroup and subpopulation | Scheduled_Table 7 | 1 | Table | Table 5 | Full analysis population |
| Disposition of patients - Patients included per geographical region and the follow-up duration | Scheduled_Table 5 | 1 | Table | Table 6 | Full analysis population |
| Disposition of patients - Excluded patients from populations | Scheduled_Listing 1 to Scheduled_Listing 3 | 1 | Listing | Listing 3 to Listing 5 | Full analysis population |
| Disposition of patients – Patient prematurely discontinued | Scheduled_Table 6 and Scheduled_Listing 4 | 1 | Table and Listing | Table 7 and Listing 6 | Full analysis population |
| Demographics and patients' characteristics | Scheduled_Table 8 | 1 & 2 | Table and Listing | Table 8 and Listing 7 | Full analysis<br>population |
| Disease history at baseline - Associated symptoms with cough | Scheduled Table 9 and Scheduled Table 10 | 182 | Table and Listing | Table 9 and Table 10 and Listing 8 | Full analysis population |
| Medical history - pre-existing medical condition | Scheduled _Table 11 | 182 | Table and Listing | Table 11 and Listing 9 | Full analysis population |
| Prior treatment for ongoing cough | Scheduled _Table 12 – 13,<br>Scheduled _Listing 5 | 1 | Listing | Listing 10 | Full analysis population |
| Ongoing concomitant treatment | Scheduled _Table 14 – 15,<br>Scheduled _Listing 6 | - | Listing | Listing 11 | Full analysis<br>population |
| All concomitant treatment during follow-up | Scheduled _Table 16 – 17,<br>Scheduled _Listing 7 | - | Listing | Listing 12 | Full analysis<br>population |
| Primary endpoint - Change in PCQ total score | Scheduled_Table 22 | 2 | Listing and patient profile | Figure 2 and Listing 13 | Performance<br>population |

| Page 14 on 81 |
|-----------------------------|
| 14/05/2025 |
| Statistical Analysis Report |
| C1735 |

| Analyses performed | Scheduled TFLs (before the premature study termination) | Based on<br>planned<br>TFLs (1) or<br>new TFLs<br>(2) | Type of TFLs to be produced | TFLs performed (after the premature study termination) | Population concerned |
|---|---|---|---|---|---|
| Secondary outcome - PCQ items | Scheduled _Table 23 to 29 | 2 | Ppatient profile | Figure 3 | Performance population |
| Secondary outcome - Daily cough severity | Scheduled_Table 30 to 33 | 2 | Listing and patient profile | Figure 4 and Listing 14 | Performance population |
| Secondary outcome - Change in PAC-QoL total score | Scheduled_Table 34 | 2 | Listing and patient profile | Figure 5 and Listing 15 | Performance<br>population |
| Secondary outcome - PAC-QoL items | Scheduled _Table 35 | 2 | Patient profile | Figure 6 | FAS population |
| Secondary outcome - Adherence | Scheduled_Table 36 | 2 | Listing | Listing 16 | FAS population |
| Secondary outcome - Satisfaction questionnaire | Scheduled_Table 37 | 1 & 2 | Table and listing | Table 12 and Listing 17 | Full analysis population |
| Secondary outcome - Summary of adverse events | Scheduled_Table 38 to 48 | 1 | Table | Table 13 (first part of the scheduled table 38, until Number of ADE per patient related to device) | Safety population |
| Secondary outcome - all AEs | Scheduled_Listing 8 to 9 | 1 | Listing | Listing 18 | Safety population |
| Secondary outcome - Device deficiencies | Scheduled_Table 49 | _ | Table | Table 14 | Safety population |

| 14/05/2025 | Page <b>15</b> on <b>81</b> |
|------------|-----------------------------|
| 11/00/2020 | i ago io on oi |

| _ | |
|----|--------|
| -c | 1721 |
| | I / 3: |

3

**Statistical Analysis Report** 

## INDEX

| 3.1 Summary Tables index | |
|---|---|
| Summary_Table 1: Analyses performed after premature study termination | 3 |
| 3.2 Tables index | |
| Table 1 : Description of Study conduct (key dates/durations) | 8256n7025573 |
| Table 13 : Adverse events – Summary of AES (SAFETY) Table 14 : Device deficiencies - SAFETY population | |
| Figure 1: Disposition of patients: Flow chart | 0<br>4<br>6<br>8<br>0<br>2<br>4<br>7<br>L |
| Figure 20 and 21: Patient profile for PAC-QoL individual items - PERFORMANCE population– item 2 of PAC-QoL | L |
| Figure 22 and 23: Patient profile for PAC-QoL individual items - PERFORMANCE population— item 3 of PAC-QoL 64 | L |
| Figure 24 and 25: Patient profile for PAC-QoL individual items - PERFORMANCE population— item 4 of PAC-QoL individual items - PERFORMANCE population— item 5 of PAC-QoL individual items - PERFORMANCE population— item 5 of PAC-QoL individual items - PERFORMANCE population— item 6 of PAC-QoL individual items - PERFORMANCE population— item | 6<br>L<br>8<br>L |
| 3.4 Listings index | |
| Listing 1: Patients not pre-selected by pharmacists* (Register 1) n=54 | 4<br>9<br>9 |

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>16</b> on <b>81</b> |
|---|---|---|---|
|---|---|---|---|

| Listing 8: Disease history – Acute dry cough diagnosis and associated symptoms at baseline – FAS popula | |
|---|---|
| (n=9) | . 36 |
| Listing 9: Medical history - Pre-existing medical conditions concomitant to cough at baseline - FAS popula | |
| (N=0) | . 38 |
| Listing 10: Prior treatment for ongoing cough at baseline -FAS population (N=1 treatment for 1 patient*) | |
| Listing 11: Ongoing concomitant treatment (other than cough treatments) at baseline - FAS population (I treatments for 2 patients) | |
| Listing 12: All concomitant treatment during follow-up – FAS population (N=2 treatments for 1 patient) | . 39 |
| Listing 13: Multi-occurrence listing (per child and per visit) for PCQ score (PERFORMANCE POPULATION) (r | 1=7)<br>. 42 |
| Listing 14: Multi-occurrence listing (per child and per visit) for VAS score (PERFORMANCE POPULATION) (n | |
| Listing 15: Multi-occurrence listing (per child and per visit) for PAC-QoL score (PERFORMANCE POPULATIOn (n=6) | (NC |
| Listing 16: Daily consumption of syrup (n=12) | . 72 |
| Listing 17: Parents' satisfaction (D3 or D4) (FAS population) (n=12 with 3 missing satisfaction questionnaires). | . 75 |
| Listing 18: Listing of all AE (n= 7 AE for 4 patients) | . 78 |

| C1735 Statistical Analysis Report | 14/05/2025 | Page <b>17</b> on <b>81</b> |
|-----------------------------------|------------|-----------------------------|
| C1/35 Statistical Analysis Report | 14/05/2025 | Page 17 on 81 |

### 4 RESULTS

The tables, figures and listings presented below are based on the database extracted on April 1st, 2025, following the database lock performed on March 31st, 2025. All content in Part 7 has been produced in accordance with the Statistical Analysis Plan, signed on March 31st, 2025.

The study spanned a period of almost 10 months, from March 9<sup>th</sup> to December 31<sup>th</sup>, 2024, corresponding to the pre-screening of the first patient and the cut-off date, given to the 45 pharmacies actively participating in the study, for inclusions, with recruitment taking place over 8 months within that period and with an effective study duration of 8-month (between March 14, 2024 and November, 7<sup>th</sup>, 2024). Remote inclusion visits were coordinated with an investigator, based at the clinical investigation site CEN Experimental, the first patient being included on March 14, 2024.

Remote follow-up of the patients lasted up to 4 days. The last patient's last visit took place on November  $7^{th}$ , 2024.

### 4.1 Description of Study Conduct

Table 1 : Description of Study conduct (key dates/durations)

| Key dates/durations at data extraction (01/04/2025) | |
|-----------------------------------------------------|------------|
| First patient in (FPI) | 14/03/2024 |
| Last patient in (LPI) | 06/11/2024 |
| Duration of inclusion period <sup>1</sup> | 8 months |
| Last patient last visit (LPLV) | 07/11/2024 |
| Duration of study <sup>2</sup> | 8 months |

<sup>&</sup>lt;sup>1</sup>Date of LPI – Date of FPI.

<sup>&</sup>lt;sup>2</sup>Date of LPLV – Date of FPI.

The recruitment was opened till 31st of December but no patient included in December

| C1735 Statistical Analysis Report | 14/05/2025 | Page <b>18</b> on <b>81</b> |
|-----------------------------------|------------|-----------------------------|
|-----------------------------------|------------|-----------------------------|

# 4.2 Children not pre-selected by pharmacists (Register 1) and not included by the investigator (Register 2)

| Number of children not pre-<br>selected by pharmacists | Parameter | N <sub>R1</sub> = 54 |
|---|---|---|
| | N | 54 |
| | Missing | 0 |
| | <6 months | 6 (11.1%) |
| Age | [6 - 12] months | 19 (35.2%) |
| | ]12 - 24] months | 16 (29.6%) |
| | ]2 - 6] years | 12 (22.2%) |
| | >6 years | 1 (1.9%) |
| Sex | N | 54 |
| | Missing | 0 |
| | Воу | 23 (42.6%) |
| | Girl | 31 (57.4%) |
| Main reasons for no | n-participation | N (%)* |
| Taking treatment(s) prof | 3 (5.6%) | |
| Associated pathology(ies) ex | 4 (7.4%) | |
| Acute dry cough | 5 (9.3%) | |
| Without prescription of the syrup for | 3 (5.6%) | |
| Refusal of parent/legal guardian | 34 (63%) | |
| Age | 7 (13%) | |
| Other rea | 3 (5.6%) | |
| Reason for refusal by parent or | | |
| Refused data of | collection | 2 (5.9%) |
| Does not have | ve time | 15 (44.1%) |
| Not interes | sted | 17 (50%) |

<sup>\*</sup>The total may exceed 100% if a patient has more than one reason for non-participation.

| Statical Analysis Donort 14/05/2005 Dono 40 cn 94 | Page <b>19</b> on <b>81</b> | /202 | Statistical Analysis Report | C1735 |
|---|---|---|---|---|
|---|---|---|---|---|

| n=54 |
|-----------------|
| $\widehat{-}$ |
| gister 1 |
| Š |
| ェ |
| harmacists* ( |
| d |
| $\overline{}$ |
| ğ |
| 0 |
| ot pre-selected |
| _ |
| $\subseteq$ |
| nts |
| atie |
| Ба |
| <u></u> |
| Υ- |
| isting |

| Dharmoniot | ל זווס ווסר ל | Designed 1. Fautelite libit pre-selected by priminacists (inclusion 1) 11-04 | Child ook | 10 11 1 100 | Dotoile of seconds I selected |
|---|---|---|---|---|---|
| riiaiiiiacist<br>ID | ٥ | (ENG) | (ENG) | Reason if other reason (ENG) | Details of parellar refusal<br>(ENG) |
| 32 | 450 | ]12 - 24]<br>months | Girl | Acute dry cough > 48 hours | |
| 32 | 454 | ]12 - 24]<br>months | Girl | Other reason: 1 single dose in the evening | |
| 32 | 466 | ]12 - 24]<br>months | Girl | Acute dry cough > 48 hours | |
| 92 | 541 | ]12 - 24]<br>months | Boy | Refusal of parent/legal guardian to participate in the study | Not interested |
| 64 | 641 | ]2 - 6] years | Boy | Refusal of parent/legal guardian to participate in the study | Does not have time |
| 88 | 693 | [6 - 12] months | Girl | Acute dry cough > 48 hours | |
| 27 | 722 | <6 months | Boy | Taking treatment(s) prohibited in the study and Age greater than 6 years old | |
| 38 | 741 | ]12 - 24]<br>months | Boy | Refusal of parent/legal guardian to participate in the study | Does not have time |
| 104 | 774 | ]12 - 24]<br>months | Boy | Refusal of parent/legal guardian to participate in the study | Does not have time |
| 92 | 777 | ]12 - 24]<br>months | Boy | Refusal of parent/legal guardian to participate in the study | Not interested |
| 104 | 780 | [6 - 12] months | Boy | Refusal of parent/legal guardian to participate in the study | Not interested |
| 92 | 812 | ]12 - 24]<br>months | Girl | Refusal of parent/legal guardian to participate in the study | Not interested |
| 104 | 833 | [6 - 12] months | Boy | Refusal of parent/legal guardian to participate in the study | Not interested |
| 92 | 841 | ]2 - 6] years | Girl | Refusal of parent/legal guardian to participate in the study | Not interested |
| 178 | 856 | [6 - 12] months | Boy | Taking treatment(s) prohibited in the study | |
| 93 | 861 | ]12 - 24]<br>months | Girl | Refusal of parent/legal guardian to participate in the study | Not interested |
| 93 | 884 | ]2 - 6] years | Boy | Taking treatment(s) prohibited in the study | |
| 42 | 915 | [6 - 12] months | Girl | Associated pathology(ies) excluded from the study | |
| 40 | 918 | ]12 - 24]<br>months | Girl | Refusal of parent/legal guardian to participate in the study | Not interested |
| 151 | 941 | ]2 - 6] years | Girl | Refusal of parent/legal guardian to participate in the study | Not interested |
| 151 | 943 | ]12 - 24]<br>months | Boy | Refusal of parent/legal guardian to participate in the study | Not interested |
| 102 | 954 | ]2 - 6] years | Girl | Refusal of parent/legal guardian to participate in the study | Does not have time |

# C1735\_RAS\_1.0\_RNSR\_20250514.docx

| Page <b>20</b> on <b>81</b> |
|-----------------------------|
| 14/05/2025 |
| Statistical Analysis Report |
| C1735 |

| Details of parental refusal (ENG) | | Does not have time | Does not have time | Does not have time | Does not have time | Not interested | Does not have time | Does not have time | Does not have time | Does not have time | | | | Not interested | Does not have time | Not interested | | Not interested | Refused data collection | Does not have time | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Reason if other reason (ENG) | Age greater than 6 years old | Refusal of parent/legal guardian to participate in the study | Refusal of parent/legal guardian to participate in the study | Refusal of parent/legal guardian to participate in the study | Refusal of parent/legal guardian to participate in the study | Refusal of parent/legal guardian to participate in the study | Refusal of parent/legal guardian to participate in the study and Age greater than 6 years old | Refusal of parent/legal guardian to participate in the study | Refusal of parent/legal guardian to participate in the study | Refusal of parent/legal guardian to participate in the study | əɓY | Associated pathology(ies) excluded from the study | Associated pathology(ies) excluded from the study | Refusal of parent/legal guardian to participate in the study | Refusal of parent/legal guardian to participate in the study | Refusal of parent/legal guardian to participate in the study | Associated pathology(ies) excluded from the study | Refusal of parent/legal guardian to participate in the study | Refusal of parent/legal guardian to participate in the study | Refusal of parent/legal guardian to participate in the study | Acute dry cough > 48 hours | Acute dry cough > 48 hours and Age greater than 6 years old | Without prescription of the syrup for an infant aged 6 to 12 months and Age greater than 6 years old |
| Child sex<br>(ENG) | Girl | Boy | Girl | Boy | Girl | Boy | Girl | Girl | Girl | Boy | Girl | Girl | Girl | Girl | Boy | Boy | Boy | Girl | Boy | Boy | Girl | Boy | Girl |
| Child age<br>(ENG) | >6 years | ]2 - 6] years | [6 - 12] months | [6 - 12] months | [6 - 12] months | [6 - 12] months | <6 months | [6 - 12] months | [6 - 12] months | [6 - 12] months | <6 months | ]12 - 24]<br>months | ]12 - 24]<br>months | [6 - 12] months | ]2 - 6] years | [6 - 12] months | ]2 - 6] years | ]2 - 6] years | ]12 - 24]<br>months | [6 - 12] months | [6 - 12] months | <6 months | <6 months |
| Child | 926 | 696 | 986 | 686 | 994 | 966 | 866 | 1004 | 1021 | 1023 | 1047 | 1075 | 1077 | 1137 | 1164 | 1166 | 1201 | 1224 | 1231 | 1243 | 1246 | 1265 | 1268 |
| Pharmacist<br>ID | 102 | 102 | 151 | 178 | 77 | 22 | 2.2 | 178 | 165 | 165 | 165 | 126 | 126 | က | 9 | 40 | 178 | 53 | 43 | 53 | 53 | 42 | 09 |

# C1735\_RAS\_1.0\_RNSR\_20250514.docx

| Page <b>21</b> on <b>81</b> |
|-----------------------------|
| 14/05/2025 |
| Statistical Analysis Report |
| C1735 |

| Pharmacist<br>ID | Child | Child age<br>(ENG) | Child sex<br>(ENG) | Reason if other reason (ENG) | Details of parental refusal (ENG) |
|---|---|---|---|---|---|
| 09 | 1272 | ]12 - 24]<br>months | Girl | Without prescription of the syrup for an infant aged 6 to 12 months | |
| 09 | 1275 | [6 - 12] months | Girl | Refusal of parent/legal guardian to participate in the study | Not interested |
| 09 | 1278 | ]12 - 24]<br>months | Boy | Refusal of parent/legal guardian to participate in the study | Not interested |
| 09 | 1280 | 1280 [6 - 12] months | Girl | Refusal of parent/legal guardian to participate in the study | Not interested |
| 38 | 1284 | 1284 [6 - 12] months | Girl | Without prescription of the syrup for an infant aged 6 to 12 months | |
| 65 | 1290 | ]2 - 6] years | Girl | Refusal of parent/legal guardian to participate in the study | Refused data collection |
| 65 | 1296 | ]2 - 6] years | Girl | Other reason: Pharmacy visit on a Saturday | |
| 53 | 1299 | <6 months | Girl | Age greater than 6 years old and Other reason: Pharmacy visit on a Saturday | |
| | | <u> </u> | | | |

<sup>\*</sup>The listing above has been sorted according to the Child ID column

**52** children referred by pharmacists were not included in the study:

- 32 for study logistics reasons:
  - o **9** out of time (weekends or after 6pm)
  - 23 parents were unreachable
- 20 children not meeting selection criteria
  - 10 are not in the ENNOV database (contacted upstream by our operators (TEC) before transmission to the PI)
    - 2 children were under 12 months of age and did not have a prescription
    - 1 child had had a cough for more than 48 hours
    - 3 children were taking or had taken a prohibited treatment in the last 15 days
    - 2 parents no longer wished to participate following a call from the investigating physician
    - 1 parent was not available for the doctor's call
    - 1 parent for whom the syrup had been dispensed 3 days before the form was completed
  - 10 are in the ENNOV database (contacted directly by the PI) (see the characteristics of the 10 children in the following tables):
    - 4 due to PCQ score criteria
    - 3 children were over 6 years old
    - 3 children were under 12 months of age and did not have a prescription

ENNOV database: number of children not included by principal investigator (after the telephone appointment): 10

The characteristics of the 10 children in the ENNOV database are described below:

Table 3 : Children not included by principal investigator (Register 2) (n=10)

| Number of children not included by principal investigator | | N <sub>R2</sub> =10 |
|---|---|---|
| Age (year) | N | 10 |
| | Missing | 0 |
| | Mean (± SD) | $4.9 \pm 4.5$ |
| | Median | 3.8 |
| | Q1-Q3 | 0.9 - 8.5 |
| | Min – Max | 0.6 - 13.8 |
| Sex | N | 10 |
| | Missing | 0 |
| | Boy | 4 (40%) |
| | Girl | 6 (60%) |
| PCQ total score before inclusion | N | 4 |
| | Missing | 6 |
| | Mean (± SD) | 8.3 ± 2.1 |
| | Median | 8.5 |
| | Q1-Q3 | 6.5 - 10 |
| | Min – Max | 6 - 10 |

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>23</b> on <b>81</b> |
|---|---|---|---|

| Do not meet eligibility criteria | N | %* Not all criteria are filled by the IP. In most cases, the IP stopped at the first criterion not met. The percentage can therefore not be presented. |
|---|---|---|
| Boys or girls aged less than 6 months or more than 6 years of age | 4 | ID103<br>ID 107<br>ID 117<br>ID 122 |
| With one of his/her parents/legal guardian having purchased Petit Drill in a pharmacy not participating in the study | 0 | |
| No confirmed prescription from a treating physician for infants between 6 months and 12 months of age | 3 | ID104<br>ID 110<br>ID 120 |
| No acute dry cough lasting less than 48 hours | 0 | |
| With a score ≥ 3 for less than 3 of the 5 PCQ questions (based on assessment the night prior to inclusion) | 4 | ID 101<br>ID 103<br>ID 119<br>ID 131 |
| No respect of the recommended daily doses* of Petit Drill during the 3 day-treatment despite child-minding None of the parents/legal guardian have a smartphone allowing using the ePRO App. NursTrial® | 0 | |
| None of the parent/legal guardian is able to understand and to complete the questionnaires | 0 | |
| No signed informed consent for the child's enrolment in the study from any parent(s)/legal guardian | 0 | |
| Presenting: | | |
| Chronic respiratory illness such as asthma, recurrent wheezing associated to viral infections and bronchitis; | | |
| Lower respiratory infections, such as bronchitis,<br>bronchiolitis, and pneumonia;<br>Tonsillitis, otitis, or sinusitis; | 0 | |
| Persistent cough lasting more than 3 weeks, whatever the etiology; | | |
| Gastrointestinal pathology, involving vomiting, nausea, or diarrhea; | | |
| With ongoing use of paracetamol, and/or homeopathic products against cough Having had corticosteroid treatment, antibiotics, | 0 | |
| antihistaminic or any cough medication (such as, but not<br>limited to, Phytoxil, Arkotoux) in the previous 15 days<br>since inclusion | 0 | |
| With a brother/sister already included in the present clinical investigation | 0 | |
| Enrolled in another clinical trial or being in a period of exclusion from a previous clinical trial. | 0 | |

<sup>\*</sup>Not all criteria were filled in by the PI. In most cases, the PI stopped at the first criterion not met. The percentage can therefore not be presented.

In bold, patient 103 for whom 2 inclusion criteria are not met

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>24</b> on <b>81</b> |
|---|---|---|---|
|---|---|---|---|

Listing 2: Patients not included by principal investigator (Register 2) (n=10)

| Patient<br>Number | Age<br>(years) | Sex | Main reasons for non-inclusion | PCQ total score before inclusion | Prescription |
|---|---|---|---|---|---|
| 6D9E.101 | 2.5 | Girl | IC5 not respected: With a score greater than 3 or equal to 3 for less than 3 of the 5 PCQ questions (based on assessment the night prior to inclusion) | 2;1;1;1;1=6 | |
| 6D9E.103 | 6.9 | Boy | IC1 not respected: Boys or girls aged less than 6 months or more than 6 years of age AND IC5 not respected: With a score greater than 3 or equal to 3 for less than 3 of the 5 PCQ questions (based on a | 2;1;1;2;1=7 | · |
| 6D9E.104 | 0.7 | Girl | IC3 not respected: No confirmed prescription from a treating physician for infants between 6 months and 12 months of age | | No |
| 6D9E.107 | 8.5 | Girl | IC1 not respected: Boys or girls aged less than 6 months or more than 6 years of age | | |
| 6D9E.110 | 0.6 | Girl | IC3 not respected: No confirmed prescription from a treating physician for infants between 6 months and 12 months of age | | No |
| 6D9E.117 | 8.9 | Boy | IC1 not respected: Boys or girls aged less than 6 months or more than 6 years of age | | |
| 6D9E.119 | 5.1 | Boy | IC5 not respected: With a score greater than 3 or equal to 3 for less than 3 of the 5 PCQ questions (based on assessment the night prior to inclusion) | 2;2;2;2=10 | |
| 6D9E.120 | 0.9 | Girl | IC3 not respected: No confirmed prescription from a treating physician for infants between 6 months and 12 months of age | | No |
| 6D9E.122 | 13.8 | Girl | IC1 not respected: Boys or girls aged less than 6 months or more than 6 years of age | | |
| 6D9E.131 | 1 | Boy | IC5 not respected: With a score greater than 3 or equal to 3 for less than 3 of the 5 PCQ questions (based on assessment the night prior to inclusion) | 2;2;2;2=10 | |

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>25</b> on <b>81</b> |
|---|---|---|---|
|---|---|---|---|

### 4.3 Disposition of patients

Table 4 : Disposition of patients – FAS population

| Table 4 : Disposition of patients – FA | | FAS population<br>N=12 |
|---|---|---|
| FAS population <sup>1</sup> | Yes | 12 |
| Reason for exclusion from the FAS population | Do not meet eligibility criteria | N=0 - 0.0% <sup>4</sup> |
| Safety population <sup>2</sup> | Yes | 12 (100%) |
| | No | 0 (0.0%) |
| If no,<br>Reason for exclusion from the<br>safety population | Children who have never taken the syrup | NA |
| Performance population <sup>3</sup> | Yes | 7 (58.3%) |
| | No | 5 (41.7%) |
| If no,<br>Reason for exclusion from the<br>performance population | Patients lost to follow-up | 0 (0.0%) |
| | Patients who discontinued the treatment | 1 (20.0%) |
| | Patients no evaluation for the primary endpoint | 0 (0.0%) |
| | Taking treatment(s) prohibited in the<br>study | 4 (80.0%) |

<sup>1</sup> Full Analysis Set (FAS) population: The analysis population will be those patients who have been included in this clinical investigation after fulfilling all selection criteria.

2 Safety population: The safety population will be made up of all patients from the FAS population who have used Petit Drill at least once.

3 Performance population: The performance population will be made up of all patients from the safety population for whom at least once evaluation of the primary outcome is available (baseline and the last assessment) and whose parent(s) or legal guardian did not withdraw their consent at any

<sup>&</sup>lt;sup>4</sup> No patients were excluded from the FAS population.

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>26</b> on <b>81</b> |
|---|---|---|---|
|---|---|---|---|

Table 5 : Subgroup and subpopulation – FAS population

| Ago oubno | mulation/ Age subgroup | All patients (FAS) |
|------------------------|------------------------|--------------------|
| Age subpo | pulation/ Age subgroup | N=12 |
| | N | 12 |
| A wa ay by a wylatia y | Missing | 0 |
| Age subpopulation | [6 months – 12 months] | 2 (16.7%) |
| | ]12 months – 6 years] | 10 (83.3%) |
| | N | 12 |
| A ma and amana | Missing | 0 |
| Age subgroup | [6 months – 24 months[ | 3 (25%) |
| | [24 months – 6 years] | 9 (75%) |

| C1735 Statistical Analysis Report 14/05/2025 | Page <b>27</b> on <b>81</b> |
|----------------------------------------------|-----------------------------|
|----------------------------------------------|-----------------------------|

Table 6 : Disposition of patients -Number of patients included per region and follow-up duration— FAS population

| | | FAS population<br>N=12 |
|---|---|---|
| Geographic region | N | 12 |
| | Missing | 0 |
| | Auvergne-Rhône-Alpes | 0 (0.0%) |
| | Bourgogne-Franche-Comté | 1 (8.3%) |
| | Bretagne | 0 (0.0%) |
| | Centre-Val de Loire | 1 (8.3%) |
| | Corse | 0 (0.0%) |
| | Grand Est | 3 (25.0%) |
| | Hauts-de-France | 2 (16.7%) |
| | Île-de-France | 0 (0.0%) |
| | Normandie | 0 (0.0%) |
| | Nouvelle-Aquitaine | 3 (25.0%) |
| | Occitanie | 2 (16.7%) |
| | Pays de la Loire | 0 (0.0%) |
| | Provence-Alpes-Côte d'Azur | 0 (0.0%) |
| Follow-up duration (days) <sup>1</sup> | N | 12 |
| | Missing | 0 |
| | Mean (± SD) | $3.6 \pm 0.8$ |
| | Median | 4 |
| | Q1-Q3 | 3.5 - 4 |
| | Min – Max | 2 - 4 |

<sup>1-</sup> Duration of study: Date of study end – Date of inclusion

Figure 1: Disposition of patients: Flow chart



| <b>al Analysis Report</b> 14/05/2025 Page <b>29</b> on <b>81</b> |
|------------------------------------------------------------------|
|------------------------------------------------------------------|

Listing 3: Patients excluded from FAS population (N=0)

| בואווווט אייר מווכוווט כאי | Figure 9. Fauerius excladed II offi 1 Ac population (14-0) | | | | | | |
|---|---|---|---|---|---|---|---|
| Patient Number | FAS population | Region | Forbidden<br>treatments at<br>inclusion | Age (years) | Sex | Reason for exclusion | Date of inclusion |
| XX-XX | No | | | | | | |
| Listing 4: Patients exc | Listing 4: Patients excluded from the Safety population $(N=0)$ | opulation (N=0) | | | | | |
| Patient Number | Safety population | Region | Forbidden<br>treatments at<br>inclusion | Age (years) | Sex | Reason for exclusion | Date of inclusion |
| XX-XX | No | | | | | | |

Listing 5: Patients excluded from the Performance population (N=5)

| -<br>- | excinded from the Pe | Isting 5. Patients excluded from the Performance population (N=5) | (C- | | | |
|---|---|---|---|---|---|---|
| Pres<br>PER<br>P | Presence of the patient in the PERFORMANCE population | Region | Age<br>calculated in<br>years | Sex<br>(D1) | Reason for exclusion from the PERFORMANCE population | Date of inclusion |
| | No | Grand Est | 1.5 | Girl | Taking treatment(s) prohibited in the study (baseline): VENTOLINE | 25/03/2024 |
| | No | Nouvelle-Aquitaine | 2.3 | Girl | Taking treatment(s) prohibited in the study (during the follow-up): CELESTENE + TUSSIDANE | 28/03/2024 |
| | No | Grand Est | 5.6 | Girl | Taking treatment(s) prohibited in the study (during the follow-up): DOLIPRANE + PIVALONE | 02/10/2024 |
| | No | Grand Est | 0.7 | Boy | Taking treatment(s) prohibited in the study (started one day before D1): DOLIPRANE | 04/11/2024 |
| | No | Hauts-de-France | 2.1 | Girl | Patient with tonsillitis: Syrup taken for only one day before diagnosis of tonsillitis (D2) Syrup taken only on the day of inclusion: D1 | 06/11/2024 |

| , | C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>30</b> on <b>81</b> |
|---|---|---|---|---|
|---|---|---|---|---|

Table 7 : Patients prematurely discontinued from the study – FAS population

| Patients prematurely discon | tinued from the study | N/% (according to FAS population) |
|---|---|---|
| Number and percentages of | Yes | 3 (25.0%) |
| patients prematurely | No | 9 (75.0%) |
| discontinued from the study | Missing | 0 |
| Reasons for premature discontinuation* | | |
| | Serious/non-serious adverse event leading to the discontinuation of Petit Drill | 1 (33.3%) |
| | Decision of parent/legal representative | 0 (0.0%) |
| | Withdrawal of consent | 0 (0.0%) |
| | Premature discontinuation of Petit Drill syrup | 1 (33.3%) |
| | Lost to follow-up | 2 (66.7%) |
| | Other reason for premature discontinuation | 0 (0.0%) |
| | Missing | 0 |

<sup>\*</sup>The total may exceed 100%, if a patient has more than one reason reasons for premature discontinuation. 3 patients and 4 reasons (patient with 2 reasons) patient 134

| Page <b>31</b> on <b>81</b> |
|-----------------------------|
| 14/05/2025 |
| Statistical Analysis Report |
| C1735 |

Listing 6: Patients who discontinued prematurely the study from FAS population (N=3)

| Subject<br>ID | Presence<br>of the<br>patient in<br>the FAS | Presence<br>of the<br>patient in<br>the<br>SAFETY | Presence of the patient in the PERFORMANCE population | Region | Treatments at<br>baseline | Age<br>calculated<br>in years | Sex | Reason for who discontinued prematurely the study | Date of<br>inclusion | Date of Date inclusion withdrawal | Follow-<br>up<br>duration<br>(days) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 6D9E.109 | | population<br>Yes | No | Grand Est | VENTOLINE | 1.5 | Girl | Lost to follow-up | 25/03/2024 | 25/03/2024 27/03/2024 | 2 |
| 6D9E.112 | Yes | Yes | Yes | Nouvelle-Aquitaine | | 3.0 | Boy | Lost to follow-up | 28/03/2024 | 28/03/2024 01/04/2024 | 4 |
| 6D9E.134 | Yes | Yes | °Z | Hauts-de-France | | 2.1 | Girl | Serious/non-serious adverse event leading to the discontinuation of Petit Drill and Premature discontinuation of Petit Drill syrup | | 06/11/2024 07/11/2024 | 7 |

<sup>1-</sup> Duration of study: Date of study end – Date of inclusion

| C1735 Statistical Analysis Report | 14/05/2025 | Page <b>32</b> on <b>81</b> |
|-----------------------------------|------------|-----------------------------|
|-----------------------------------|------------|-----------------------------|

## 4.4 Clinical and sociodemographic characteristics of children using Petit Drill (FAS population)

### 4.4.1 Baseline demographics (FAS population)

Table 8: Demographic and patient's characteristics at baseline – FAS population

| | | All patients (FAS |
|--------------------------|------------------------|-------------------|
| | | N=12 |
| | N | 12 |
| | Missing | 0 |
| A 1 () | Mean (± SD) | 3.1 ± 1.9 |
| Age <sup>1</sup> (years) | Median | 2.7 |
| | Q1-Q3 | 1.8 - 4.8 |
| | Min – Max | 0.7 - 6 |
| | N | 12 |
| | Missing | 0 |
| | Mean (± SD) | 37.6 ± 22.4 |
| Age (months) | Median | 31.9 |
| | Q1-Q3 | 22 - 57.7 |
| | Min – Max | 8.1 - 71.7 |
| | N | 12 |
| | Missing | 0 |
| Age subgroup | [6 months – 24 months[ | 3 (25%) |
| | [24 months – 6 years] | 9 (75%) |
| | N | 12 |
| _ | Missing | 0 |
| Sex | Воу | 5 (41.7%) |
| | Girl | 7 (58.3%) |
| | N | 12 |
| | Missing | 0 |
| W | Mean (± SD) | 15.5 ± 4.2 |
| Weight (kg) | Median | 13.8 |
| | Q1-Q3 | 12.5 - 20 |
| | Min – Max | 9.9 - 22 |
| | N | 12 |
| | Missing | 0 |
| Hadada A | Mean (± SD) | 96.9 ± 13.8 |
| Height (cm) | Median | 95 |
| | Q1-Q3 | 87.5 - 107 |
| | Min – Max | 75 - 120 |

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>33</b> on <b>81</b> |
|---|---|---|---|
| | | N | 12 |
| | | Missing | 0 |
| | | Thinness | 0 (0.0%) |
| | | Normal | 11 (91.7%) |
| | | Overweight | 1 (8.3%) |
| PMI / | (kg/m²)² ———— | Obese | 0 (0.0%) |
| DIVII ( | kg/iii ) | N | 12 |
| | | Missing | 0 |
| | | Mean (± SD) | 16.4 ± 1.6 |
| | | Median | 16.3 |
| | | Q1-Q3 | 15.5 - 17.5 |
| | | Min – Max | 13.8 - 19.2 |
| | | N | 12 |
| | | Missing | 0 |
| Total number | of children in the | Mean (± SD) | 2.1 ± 0.9 |
| | (siblings) | Median | 2 |
| | | Q1-Q3 | 1.5 - 2.5 |
| | | Min – Max | 1 - 4 |
| | | N | 12 |
| | | Missing | 0 |
| | | Only child | 3 (25%) |
| Rank amo | ong siblings | 1 | 4 (33.3%) |
| | | 2 | 2 (16.7%) |
| | | 3 | 2 (16.7%) |
| | | 4 and + | 1 (8.3%) |

<sup>1 –</sup> Age: Date of inclusion – Date of Birth. 2 – BMI: calculating with the corpulence diagram

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>34</b> on <b>81</b> |
|---|---|---|---|

Listing 7: Demographic and patient's characteristics at baseline – FAS population (n=12)

| Presence of the of the patient in patient in the the PERFORMANCE SAFETY population | Da<br>incl. | Date of calc | Age<br>calculated<br>in years | Age subgroup | Sex | Weight | Height | Body<br>mass<br>index (in<br>classes) | Number of<br>children in<br>the family<br>(Siblings) | Rank<br>among<br>siblings |
|---|---|---|---|---|---|---|---|---|---|---|
| Yes Yes Hauts-de-France | | 14/03/2024 | 5.3 | [24 months – 6 years] | Girl | 21 | 117 | Normal | 2 | - |
| Yes No Grand Est | 25/0、 | 25/03/2024 | 1.5 | [6 months - 24 months] | Girl | 14 | 88 | Normal | 3 | က |
| Yes No Nouvelle-Aquitair | e( | 28/03/2024 | 2.3 | [24 months – 6 years] | Girl | 13 | 97 | Normal | 4 | 4 and<br>more |
| Yes Yes Nouvelle-Aquitaine | | 28/03/2024 | 3.0 | [24 months – 6 years] | Boy | 12 | 87 | Normal | 2 | _ |
| Yes Yes Nouvelle-Aquitai | ne | 28/03/2024 | 4.3 | [24 months – 6 years] | Boy | 22 | 107 | Overweight | 2 | 1 |
| Yes Yes Centre-Val de Loire | | 29/03/2024 | 3.9 | [24 months – 6 years] | Girl | 16 | 100 | Normal | 2 | 1 |
| Yes Yes Occitanie | 03/0. | 03/04/2024 | 0.7 | [6 months - 24 months[ | Boy | 11.4 | 82 | Normal | 7 | Only |
| Yes Yes Bourgogne-Franche- | Comté | 04/04/2024 | 0.9 | [24 months – 6 years] | Girl | 20 | 107 | Normal | 3 | 3 |
| Yes No Grand Est | | 02/10/2024 | 5.6 | [24 months – 6 years] | Girl | 20 | 120 | Normal | 2 | 2 |
| Yes Yes Occitanie | | 14/10/2024 | 2.2 | [24 months – 6 years] | Boy | 13.5 | 06 | Normal | 2 | 2 |
| Yes No Grand Est | | 04/11/2024 | 0.7 | [6 months - 24 months[ | Boy | 6.6 | 75 | Normal | 1 | Only |
| Yes No Hauts-de-France | | 06/11/2024 | 2.1 | [24 months – 6 years] | Girl | 13.5 | 93 | Normal | _ | Only |

### 4.4.2 Disease history at baseline (FAS population)

Table 9 : Acute dry cough diagnosis - FAS population

| | | FAS Population<br>(N=12) |
|---|---|---|
| | N | 12 |
| | Missing | 0 |
| Acute dry cough diagnosis: Time between | Mean (± SD) | 1.5 ± 0.7 |
| date of onset of acute dry cough symptoms<br>and date of inclusion (days) | Median | 2 |
| | Q1-Q3 | 1 - 2 |
| | Min – Max | 0 - 2 |
| Acute duy cough dispussion in cotonovice | < 1 day | 1 (8.3%) |
| Acute dry cough diagnosis in categories | [1 – 2 days] | 11 (91.7%) |

| able 10 : Associated symptoms with cough at b | | FAS Population (N=12) |
|---|---|---|
| | N | 12 |
| Patients with at least one associated<br>symptom with cough | No | 3 (25%) |
| ., , | Yes | 9 (75%) |
| | N | 9 |
| | Missing | 0 |
| N | Mean (± SD) | 1.4 ± 0.7 |
| Number of associated symptoms with cough | Median | 1 |
| | Q1-Q3 | 1 - 1 |
| | Min – Max | -1 - 3 |
| | N | 9 |
| | Missing | 0 |
| Number of associated symptoms with cough | 0 | 0 (0.0%) |
| in category | 1 | 6 (66.7%) |
| | 2 | 2 (22.2%) |
| | Missing Mean (± SD) Median Q1-Q3 Min − Max N Missing 0 1 2 ≥3 N Missing Fever Runny nose Congestion h* Sore throat Ear pain Other sensation of pain (which may be expressed in younger children by crying more | 1 (11.1%) |
| | N | 9 |
| | Missing | 0 |
| | Fever | 0 (0.0%) |
| | Runny nose | 8 (88.9%) |
| | Congestion | 1 (11.1%) |
| Type of associated symptoms with cough* | Sore throat | 2 (22.2%) |
| | Ear pain | 0 (0.0%) |
| | | 1 (11.1%) |
| | Digestive symptoms (vomiting or diarrhea) | 0 (0.0%) |
| | Reduced appetite | 1 (11.1%) |

<sup>\*</sup>The total may exceed 100%, if a patient has more than one associated symptom with cough

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>36</b> on <b>81</b> |
|---|---|---|---|

Listing 8: Disease history – Acute dry cough diagnosis and associated symptoms at baseline – FAS population (n=9)

| Presence of | Presence of | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of the | Presence of

| 5 | | | The second secon | | (1) | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Presence of<br>the patient in<br>the FAS<br>population | Presence of<br>the patient in<br>the SAFETY<br>population | Presence of the patient in the PERFORMANCE population | Region | Date of inclusion | Age<br>calculated in<br>years | Sex | Start date of dry cough | Combined associated symptoms at baseline |
| 6D9E.109 | Yes | səA | No | Grand Est | 25/03/2024 | 1.5 | Girl | 23/03/2024 | Runny nose |
| 6D9E.111 | Yes | Yes | ON. | Nouvelle-Aquitaine | 28/03/2024 | 2.3 | Girl | 27/03/2024 | Runny nose<br>+Sore throat<br>+Reduced<br>appetite |
| 6D9E.113 | Yes | səA | Yes | Nouvelle-Aquitaine | 28/03/2024 | 4.3 | Boy | 27/03/2024 | Runny nose |
| 6D9E.114 | Yes | Yes | Yes | Centre-Val de Loire | 29/03/2024 | 3.9 | Girl | 27/03/2024 | Runny nose<br>+Other sensation<br>of pain |
| 6D9E.118 | Yes | səA | Yes | Bourgogne-Franche-Comté | 04/04/2024 | 0.9 | Girl | 03/04/2024 | Runny nose |
| 6D9E.127 | Yes | Yes | No | Grand Est | 02/10/2024 | 5.6 | Girl | 30/09/2024 | Runny nose<br>+Sore throat |
| 6D9E.129 | Yes | Yes | Yes | Occitanie | 14/10/2024 | 2.2 | Boy | 12/10/2024 | Runny nose |
| 6D9E.133 | Yes | Yes | No | Grand Est | 04/11/2024 | 0.7 | Boy | 04/11/2024 | Congestion |
| 6D9E.134 | Yes | Yes | No | Hauts-de-France | 06/11/2024 | 2.1 | Girl | 04/11/2024 | Runny nose |
| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>37</b> on <b>81</b> |
|---|---|---|---|
|---|---|---|---|

### 4.4.3 Medical history at baseline (FAS population)

Table 11 : Pre-existing medical conditions concomitant to cough at baseline – FAS population

| able 11. Fre-existing medical conditions concomit | | FAS Population<br>(N=12) |
|---|---|---|
| | N | 12 |
| Patients with at least one pre-existing medical | Missing | 0 |
| condition concomitant to cough | No | 12 (100%) |
| | Yes | 0 (0.0%) |
| | N | 12 |
| | Missing | 0 |
| Niverbourge and acceptance and an acceptance | Mean (± SD) | 0 |
| Number of pre-existing medical conditions | Median | 0 |
| | Q1-Q3 | 0 - 0 |
| | Min – Max | 0 - 0 |
| | N | 12 |
| | Missing | 0 |
| Number of pre-existing medical conditions in | 0 | 12 (100%) |
| category | 1 | 0 (0.0%) |
| | 2 | 0 (0.0%) |
| | ≥3 | 0 (0.0%) |
| | N | 12 |
| | Missing | 0 |
| | Asthma | 0 (0.0%) |
| | Bronchitis | 0 (0.0%) |
| | Bronchiolitis | 0 (0.0%) |
| | Pneumonia | 0 (0.0%) |
| Type of pre-existing medical conditions | Tonsillitis | 0 (0.0%) |
| | Otitis | 0 (0.0%) |
| | Sinusitis | 0 (0.0%) |
| | Vomiting | 0 (0.0%) |
| | Nausea | 0 (0.0%) |
| | Diarrhea | 0 (0.0%) |
| | Other | 0 (0.0%) |

| C1735 Statistical Analysis Report 14/05/2025 | Page <b>38</b> on <b>81</b> |
|---|---|
|---|---|

Listing 9: Medical history – Pre-existing medical conditions concomitant to cough at baseline – FAS population (N=0)

| Patient<br>Number | FAS population | Safety<br>population | Performance<br>population | Region | Date of inclusion | Age (years) | Sex | Date of<br>acute dry<br>cough | Type of pre-existing medical conditions |
|---|---|---|---|---|---|---|---|---|---|
| XX-XX | Yes | | | | | | | | |

## 4.4.4 Prior treatment for ongoing cough at baseline (FAS population)

Listing 10: Prior treatment for ongoing cough at baseline -FAS population (N=1 treatment for 1 patient\*)

| Duration of concomitta nt medication (day) | 1 |
|---|---|
| End date | Inhalatio 25/03/202 26/03/202 n 4 |
| Route Start date End date | 25/03/202<br>4 |
| Route | Inhalatio<br>n |
| Frequenc R | Once<br>daily |
| er e | hG |
| Unit | Othe |
| Dos | ETA- Othe µG EPT 100 r |
| Anatomical ATC classification Dos Unit on mame | RESPIRATOR 2-<br>Y SYSTEM ADRENORECEPT OR AGONISTS |
| Anatomical<br>group | RESPIRATOR<br>Y SYSTEM |
| Date of Treatment Drug name inclusion | 25/03/202 VENTOLIN VENTOLINE R. SALBUTAMO |
| Treatment | VENTOLIN<br>E |
| Date of inclusion | 25/03/202<br>4 |
| Sex | 1.5 Girl |
| Ag | 1.5 |
| FA Safet Performanc Ag<br>S y e e | o<br>Z |
| Safet<br>y | Yes |
| A s | Yes |
| Subject ID | 6D9E.109 Yes Yes |
| L | L |

<sup>\*</sup> Ventoline treatment was entered into the database by the principal investigator as a treatment for cough, but without specifying its indication. At the time of data review, this treatment be a treatment without indication, without specifying whether it was a treatment for current cough or for another reason.

# 4.4.5 Ongoing concomitant treatment (other than cough treatments) at baseline (FAS population)

Listing 11: Ongoing concomitant treatment (other than cough treatments) at baseline - FAS population (N=3 treatments for 2 patients)

| т | 3 |
|---|---|
| 05/10/20 | 07/11/20<br>24 |
| 02/10/20 | 03/11/20 07/11/20<br>24 24 |
| Other | Oral |
| 1 time<br>only | Twice<br>daily |
| PULVERISATI<br>ON | Other DOSE/POIDS |
| Other | Other |
| - | - |
| CORTICOSTEROI<br>DS ACTING<br>LOCALLY | ANILIDES |
| V III Z | NERVOUS<br>SYSTEM |
| | DOLIPRA<br>NE |
| PIVALONE | DOLIPRA<br>NE |
| 02/10/20 | 04/11/20<br>24 |
| Girl | Boy |
| 5.6 | 0.7 |
| o <sub>N</sub> | No |
| Yes | 6D9E.133 Yes Yes |
| Yes | Yes |
| 127 | E. 133 |
| | 5.6 Girl 224 PIVALONE RY TRACT CORTICOSTEROI DS ACTING 1 Other ON ON ON SM SM |

| C1735 Statistical Analysis Report 14/05/2025 Page 39 on 81 |
|------------------------------------------------------------|

## 4.5 Concomitant treatments during follow up (FAS population)

Listing 12: All concomitant treatment during follow-up – FAS population (N=2 treatments for 1 patient)

| ı | r fa | | |
|---|---|---|---|
| | Duration of concomitta nt medication (day) | ဇ | 8 |
| | End date | 31/03/20<br>24 | 31/03/20<br>24 |
| | Start<br>date | Oral 30/03/20 31/03/20 | 30/03/20 31/03/20<br>24 24 |
| | Rout<br>e | Oral | Oral |
| | Frequen Rout | 1 time<br>only | 1 time<br>only |
| | Other<br>unite | | CUILLER<br>E<br>MESURE |
| | Unit | Drop | Othe |
| | n Dos Unit | 70 | 1 |
| ויין, | ATC classification<br>name | ALIMENTARY CORTICOSTEROIDS TRACT AND FOR LOCAL ORAL 70 METABOLISM TREATMENT | ESPIRATORY OPIUM ALKALOIDS SYSTEM AND DERIVATIVES |
| יישן י וטו טווטוווי | Anatomical<br>group | ALIMENTARY<br>TRACT AND<br>METABOLISM | RESPIRATORY<br>SYSTEM |
| Figure 12:7 in concommant treatment against the population (12 the particular) | Drug name | CELESTENE / [BETAMETHASO NE] | TUSSIDANE |
| מסק כיי | Indicati<br>on | TOUX | TOUX |
| י שה ייכוו | Treatment | 2.3 Girl 28/03/20 CELESTE TG | 2.3 Girl 28/03/20 TUSSIDAN TG |
| r adiii igi ic | Date of<br>inclusio<br>n | 28/03/20<br>24 | 28/03/20<br>24 |
| | S <sub>e</sub> × | Girl | Girl |
| 5 | Ag | 2.3 | 2.3 |
| יוויייי | Performan<br>ce | <sub>S</sub> | No |
| 5 | Safet<br>y | Yes | Yes |
| 9 | S S | Yes | Yes |
| FISH | Subject ID FA Safet Performan Ag Se inclusio Treatment Ce x n | 6D9E.111 Yes Yes | 6D9E.111 Yes Yes |

### 4.6 Primary endpoint - Change in PCQ total score (PERFORMANCE POPULATION)

Figure 2 and 3: Patient profile for PCQ total score - PERFORMANCE population





| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>42</b> on <b>81</b> |
|---|---|---|---|

Patients with a 3-point decrease

Delta between baseline and each day

> PCQ Score

Yes

4 42

4 6 5

15

Yes

6- 4-

15 10 25 16 Yes

7

-9

Yes

-13

6 2 5

15 12 17

-10

e e o

3

Yes

7

Not at all Somewhat

Occasionally

Not at all

Not at all

Occasionally

Boy

- 9 9 9 9

06/04/2024

03/04/2024 04/04/2024 04/04/2024

X es Kes

Yes

Yes Yes Yes

DAY 4

6D9E.116

Somewhat

A little

A little

Somewhat

G G G

04/04/2024

05/04/2024

Yes

DAY 2

6D9E.118

DAY 1

6D9E.118

Yes

DAY 3 DAY 4

6D9E.118

6D9E.118

Yes

04/04/2024

Yes

4

Occasionally Occasionally
Occasionally

Occasionally Occasionally

Girl

07/04/2024

Yes

9 1- 6

**~** 9

Occasionally | Occasionally

Occasionally

A little A little

A little

Not at all

A little

73

Occasionally Occasionally Occasionally Somewhat Somewhat Somewhat Extremely Extremely Somewhat Somewhat Somewhat Somewhat Not at all Not at all Not at all A little A little Q5 Occasionally Occasionally Occasionally Somewhat Somewhat Somewhat Somewhat Somewhat Somewhat Very much Extremely Extremely Not at all A little A little A little A little 8 Occasionally Somewhat Somewhat Somewhat Somewhat Very much Extremely Extremely Not at all Not at all Not at all Not at all Not at all A little A little A little A little ဗ Listing 13: Multi-occurrence listing (per child and per visit) for PCQ score (PERFORMANCE POPULATION) (n=7) Occasionally Occasionally Somewhat Somewhat Very much Somewhat Somewhat Extremely Extremely Not at all Not at all Not at all Not at all A little A little A little A little 8 Occasionally Occasionally Occasionally Occasionally Somewhat Very much Somewhat Very much Somewhat Somewhat Somewhat Somewhat Somewhat Extremely Not at all A little A little ð Girl Boy Girl Boy Boy Boy Boy Boy Ğij Sex Girl Boy Boy Boy Ģ Girl Girl Ģ 4 4 4 4 4 4 \_ \_ Age 4 \_ 2 က 2 2 2 က က Questionnaire Date 29/03/2024 30/03/2024 31/03/2024 01/04/2024 03/04/2024 04/04/2024 29/03/2024 30/03/2024 05/04/2024 15/03/2024 16/03/2024 17/03/2024 29/03/2024 30/03/2024 31/03/2024 28/03/2024 14/03/2024 Inclusion Date 29/03/2024 29/03/2024 03/04/2024 03/04/2024 03/04/2024 14/03/2024 14/03/2024 14/03/2024 14/03/2024 28/03/2024 28/03/2024 28/03/2024 28/03/2024 28/03/2024 28/03/2024 29/03/2024 29/03/2024 Performance population Yes Safety population Yes FAS population Yes Visit number DAY 2 DAY3 DAY 2 DAY3 DAY3 DAY 1 DAY 2 DAY3 DAY 4 DAY3 DAY 2 DAY 4 DAY 2 DAY 1 DAY 1 DAY 1 DAY 1 6D9E.116 6D9E.116 6D9E.116 6D9E.112 6D9E.112 6D9E.112 6D9E.114 6D9E.102 6D9E.102 6D9E.102 6D9E.113 6D9E.113 6D9E.113 6D9E.114 6D9E.114 6D9E.114 6D9E.102 Patient number

### C1735\_RAS\_1.0\_RNSR\_20250514.docx

| Page <b>43</b> on <b>81</b> |
|-----------------------------|
| 14/05/2025 |
| Statistical Analysis Report |
| C1735 |

| t 3- | | |
|---|---|---|
| Patients<br>with a 3-<br>point<br>decrease | | Yes |
| Delta<br>between<br>baseline<br>and<br>each<br>day | | -16 |
| PCQ<br>Score | 18 | 2 |
| Q5 | Very much | Not at all |
| 90 | Very much | Occasionally Not at all |
| 83 | Somewhat | Not at all |
| 02 | Very much Somewhat Very much | Not at all |
| 9 | Somewhat | 2 Boy Occasionally Not at all |
| Sex | 2 Boy | Boy |
| Age Sex | 2 | 2 |
| Questionnaire<br>Date | 14/10/2024 | 15/10/2024 |
| Inclusion<br>Date | 14/10/2024 | 14/10/2024 |
| Visit FAS Safety Performance number population | Yes | Yes |
| Safety<br>population | Yes | Yes |
| FAS | Yes | Yes |
| Visit | DAY 1 | DAY 2 |
| Patient<br>number | 6D9E.129 DAY 1 | 6D9E.129 DAY 2 |

PCQ. Q1. Cough frequency the night before the first syrup intake: "Q1. How frequent was your child's cough last night?"

PCQ. Q2. Sleep disturbance of the child the night before the first syrup intake: "Q2. How much did last night's cough affect your child's ability to sleep?"

PCQ. Q3. Sleep disturbance of the parent the night before the first syrup intake: "Q3. How much did last night's cough affect your ability to sleep?"

PCQ. Q4. Cough severity the night before the first syrup intake: "Q4. How severe was your child's cough last night?"

PCQ. Q5. Degree of bothersomeness to the child the night before the first syrup intake: "Q5. How bothersome was last night's cough to your child?"

### 4.7 Secondary outcome - PCQ items (PERFORMANCE POPULATION)





















Figure 12 and 13: Patient profile for PCQ items - PERFORMANCE population - item 5 of PCQ





### 4.8 Secondary outcome - Daily cough severity (VAS) (PERFORMANCE POPULATION\*)

\* This analysis was carried out on the Performance population but without patient 112, who could not be assessed at baseline.

Figure 14 and 15: Patient profile for VAS score - PERFORMANCE population





| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>56</b> on <b>81</b> |
|---|---|---|---|

Listing 14: Multi-occurrence listing (per child and per visit) for VAS score (PERFORMANCE POPULATION) (n=6)

| g<br>q | | | | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Delta between<br>baseline and<br>each day | • | -15 | -44 | -55 | - | -21 | -80 | - | -26 | -25 | -39 | • | 2 | -29 | -41 | - | 5 | -14 | -17 | • | 2 |
| VAS Score | 99 | 51 | 22 | 11 | 26 | 9/ | 17 | 20 | 24 | 25 | 11 | 99 | 28 | 27 | 15 | 38 | 43 | 24 | 21 | 6 | 11 |
| Sex | Girl | Girl | Girl | Girl | Boy | Boy | Boy | Girl | Girl | Girl | Girl | Boy | Boy | Boy | Boy | Girl | Girl | Girl | Girl | Boy | Boy |
| Age | 5.3 | 5.3 | 5.3 | 5.3 | 4.3 | 4.3 | 4.3 | 3.9 | 3.9 | 3.9 | 3.9 | 0.7 | 0.7 | 0.7 | 0.7 | 9 | 9 | 9 | 9 | 2.2 | 2.2 |
| Questionnaire Date | 14/03/2024 | 15/03/2024 | 16/03/2024 | 17/03/2024 | 28/03/2024 | 29/03/2024 | 30/03/2024 | 29/03/2024 | 30/03/2024 | 31/03/2024 | 01/04/2024 | 03/04/2024 | 04/04/2024 | 05/04/2024 | 06/04/2024 | 04/04/2024 | 05/04/2024 | 06/04/2024 | 07/04/2024 | 14/10/2024 | 15/10/2024 |
| Inclusion Date | 14/03/2024 | 14/03/2024 | 14/03/2024 | 14/03/2024 | 28/03/2024 | 28/03/2024 | 28/03/2024 | 29/03/2024 | 29/03/2024 | 29/03/2024 | 29/03/2024 | 03/04/2024 | 03/04/2024 | 03/04/2024 | 03/04/2024 | 04/04/2024 | 04/04/2024 | 04/04/2024 | 04/04/2024 | 14/10/2024 | 14/10/2024 |
| Performance population | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| Safety<br>population | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| FAS population | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| Visit number | DAY 1 | DAY 2 | DAY3 | DAY 4 | DAY 1 | DAY 2 | DAY3 | DAY 1 | DAY 2 | DAY3 | DAY 4 | DAY 1 | DAY 2 | DAY3 | DAY 4 | DAY 1 | DAY 2 | DAY3 | DAY 4 | DAY 1 | DAY 2 |
| Patient number | 6D9E.102 | 6D9E.102 | 6D9E.102 | 6D9E.102 | 6D9E.113 | 6D9E.113 | 6D9E.113 | 6D9E.114 | 6D9E.114 | 6D9E.114 | 6D9E.114 | 6D9E.116 | 6D9E.116 | 6D9E.116 | 6D9E.116 | 6D9E.118 | 6D9E.118 | 6D9E.118 | 6D9E.118 | 6D9E.129 | 6D9E.129 |

### 4.9 Secondary outcome - Change in PAC-QoL total score\*

\* This analysis was carried out on the Performance population but without patient 112, who could not be assessed at baseline.

Figure 16 and 17: Patient profile for PAC-QoL total score - PERFORMANCE population





| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>59</b> on <b>81</b> |
|---|---|---|---|

Listing 15: Multi-occurrence listing (per child and per visit) for PAC-QoL score (PERFORMANCE POPULATION) (n=6)

| ne r | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Delta<br>between<br>baseline<br>and<br>each<br>day | | 0.17 | | 2.83 | | 0 | | -0.5 | | 1 | | 0 |
| PAC-<br>QoL<br>Score | 4 | 4.2 | 3.5 | 6.3 | 5.3 | 5.3 | 9 | 5.5 | 5.2 | 6.2 | 4.3 | 4.3 |
| 90 | None of<br>the time | None of<br>the time | None of<br>the time | None of<br>the time | None of<br>the time | None of<br>the time | None of<br>the time | None of<br>the time | Hardly<br>any of<br>the time | None of<br>the time | Some of<br>the time | Once in<br>a while |
| 90 | Very worried /<br>concerned | Fairly worried /<br>concerned | Somewhat<br>worried /<br>concerned | A little worried / concerned | Fairly worried / concerned | Very worried / concerned | A little worried /<br>concerned | A little worried / concerned | Somewhat<br>worried /<br>concerned | A little worried /<br>concerned | Fairly worried /<br>concerned | Somewhat<br>worried /<br>concerned |
| Q4 | Somewhat<br>worried /<br>concerned | Somewhat<br>worried /<br>concerned | Fairly worried / concerned | Not worried /<br>concerned | Hardly worried / concerned | Not worried /<br>concerned | Hardly worried / concerned | A little worried / concerned | A little worried / concerned | Hardly worried /<br>concerned | Somewhat<br>worried /<br>concerned | A little worried / concerned |
| Q3 | Very worried /<br>concerned | Somewhat<br>worried /<br>concerned | Fairly worried /<br>concerned | Not worried /<br>concerned | Hardly worried / concerned | A little worried / concerned | Hardly worried /<br>concerned | Hardly worried / concerned | A little worried /<br>concerned | Hardly worried /<br>concerned | Somewhat<br>worried /<br>concerned | Somewhat<br>worried /<br>concerned |
| 02 | Hardly<br>any of<br>the time | Some of<br>the time | Most of<br>the time | Once in<br>a while | Some of<br>the time | Some of<br>the time | Hardly<br>any of<br>the time | Some of<br>the time | Hardly<br>any of<br>the time | Hardly<br>any of<br>the time | Some of<br>the time | Some of<br>the time |
| Q1 | Fairly worried / concerned | Fairly worried / concerned | Very worried /<br>concerned | Not worried /<br>concerned | Hardly worried / concerned | Not worried /<br>concerned | Hardly worried<br>/ concerned | Hardly worried / concerned | A little worried /<br>concerned | Not worried /<br>concerned | Not worried /<br>concerned | Somewhat<br>worried /<br>concerned |
| Sex | Girl | Girl | Boy | Boy | Girl | Girl | Boy | Boy | Girl | Girl | Boy | Boy |
| Age | 5.3 | 5.3 | 4.3 | 4.3 | 3.9 | 3.9 | 0.7 | 0.7 | 9 | 9 | 2.2 | 2.2 |
| Questionnaire<br>Date | 14/03/2024 | 17/03/2024 | 28/03/2024 | 31/03/2024 | 29/03/2024 | 01/04/2024 | 03/04/2024 | 06/04/2024 | 04/04/2024 | 07/04/2024 | 14/10/2024 | 16/10/2024 |
| Inclusion<br>Date | 14/03/2024 | 14/03/2024 | 28/03/2024 | 28/03/2024 | 29/03/2024 | 29/03/2024 | 03/04/2024 | 03/04/2024 | 04/04/2024 | 04/04/2024 | 14/10/2024 | 14/10/2024 |
| Performance<br>population | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| Safety<br>population | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| FAS<br>population | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes | Yes |
| Visit<br>number | DAY 1 | DAY 4 | DAY 1 | DAY 4 | DAY 1 | DAY 4 | DAY 1 | DAY 4 | DAY 1 | DAY 4 | DAY 1 | DAY 3 |
| Patient<br>number | 6D9E.102 | 6D9E.102 | 6D9E.113 | 6D9E.113 | 6D9E.114 | 6D9E.114 | 6D9E.116 | 6D9E.116 | 6D9E.118 | 6D9E.118 | 6D9E.129 | 6D9E.129 |

Q1. Worried and/or concerned about the child's cough getting worse Q2. Feeling tired and/or exhausted because of the child's cough Q3. Worried/concerned about the effects of your child's cough on him/her Q4. Worried and/or concerned about the cause of the child's cough Q5. Worried and/or concerned that the child didn't sleep well due to cough Q6. Change in family commitments due to child's cough

### 4.10 Secondary outcome - PAC-QoL items\*

Figure 18 and 19: Patient profile for PAC-QoL individual items - PERFORMANCE population- item 1 of PAC-QoL



<sup>\*</sup> This analysis was carried out on the Performance population but without patient 112, who could not be assessed at baseline.



| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>62</b> on <b>81</b> |
|---|---|---|---|
|---|---|---|---|

Figure 20 and 21: Patient profile for PAC-QoL individual items - PERFORMANCE population- item 2 of PAC-QoL





Figure 22 and 23: Patient profile for PAC-QoL individual items - PERFORMANCE population- item 3 of PAC-QoL





Figure 24 and 25: Patient profile for PAC-QoL individual items - PERFORMANCE population- item 4 of PAC-QoL



**Statistical Analysis Report** 



| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>68</b> on <b>81</b> |
|---|---|---|---|
|---|---|---|---|

Figure 26 and 27: Patient profile for PAC-QoL individual items - PERFORMANCE population- item 5 of PAC-QoL





Figure 28 and 29: Patient profile for PAC-QoL individual items - PERFORMANCE population- item 6 of PAC-QoL





| Page <b>72</b> on <b>81</b> |
|-----------------------------|
| 14/05/2025 |
| Statistical Analysis Report |
| C1735 |

### 4.11 Secondary outcome - Adherence (FAS population)

Listing 16: Daily consumption of syrup (n=12)

| Patient<br>number | FAS<br>population | Safety<br>population | Performance<br>population | Inclusion<br>Date | Age | Sex | Nb<br>dose<br>D1 | Syrup<br>taken the<br>day before<br>D2 | Nb<br>dose<br>D2 | Syrup<br>taken the<br>day before<br>D3 | Nb<br>dose<br>D3 | Syrup<br>taken the<br>day before<br>D4 | Nb<br>dose<br>D4 | Nb<br>dose<br>D5 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 6D9E.102 | Yes | Yes | Yes | 14/03/2024 | 5.3 | Girl | 2 | ХeУ | 3 | Yes | _ | Yes | 3 | 0 |
| 6D9E.109 | Yes | Yes | No | 25/03/2024 | 1.5 | Girl | 0 | ХeУ | 0 | | 0 | | 0 | 0 |
| 6D9E.111 | Yes | Yes | No | 28/03/2024 | 2.3 | Girl | 1 | Yes | 4 | Yes | 4 | Yes | 2 | 0 |
| 6D9E.112 | Yes | Yes | Yes | 28/03/2024 | 3 | Boy | 0 | ХəУ | 0 | Yes | 0 | | 0 | 0 |
| 6D9E.113 | Yes | Yes | Yes | 28/03/2024 | 4.3 | Boy | 0 | ХeУ | 2 | Yes | 0 | No | 0 | 0 |
| 6D9E.114 | Yes | Yes | Yes | 29/03/2024 | 3.9 | Girl | 2 | Yes | 3 | Yes | 3 | Yes | 2 | 1 |
| 6D9E.116 | Yes | Yes | Yes | 03/04/2024 | 0.7 | Boy | 1 | ХeУ | 3 | Yes | 2 | Yes | 1 | 0 |
| 6D9E.118 | Yes | Yes | Yes | 04/04/2024 | 9 | Girl | 1 | Yes | 3 | Yes | 3 | Yes | 1 | 0 |
| 6D9E.127 | Yes | Yes | No | 02/10/2024 | 5.6 | Girl | 1 | Yes | 3 | Yes | 2 | Yes | 3 | 0 |
| 6D9E.129 | Yes | Yes | Yes | 14/10/2024 | 2.2 | Boy | 1 | Yes | 2 | No | 0 | | 0 | 0 |
| 6D9E.133 | Yes | Yes | No | 04/11/2024 | 0.7 | Boy | 0 | Yes | 3 | Yes | 2 | Yes | 2 | 0 |
| 6D9E.134 | səД | Yes | oN | 06/11/2024 | 2.1 | Girl | 0 | ХeУ | 0 | | 0 | | 0 | 0 |

| 14/05/2025 | Page <b>73</b> on <b>81</b> |
|------------|-----------------------------|
|------------|-----------------------------|

### 4.12 Secondary outcome - Satisfaction questionnaire (FAS population)

Table 12: Parents' satisfaction with Petit Drill, at 2-day treatment or at 3-day treatment - FAS population

| | Satisfaction — | ay treatment – FAS population All patients (FAS population) N=12 |
|---|---|---|
| | | D4 n= 8 (or D3 n=1)* |
| | N | 9 |
| | Missing | 3 |
| Quality of therapeutic | Excellent | 2 (22.2%) |
| nanagement received by<br>the child | Good | 5 (55.6%) |
| | Fair | 1 (11.1%) |
| | Poor | 1 (11.1%) |
| | N | 9 |
| | Missing | 3 |
| Response to the child's | Almost all my child's needs were met | 2 (22.2%) |
| needs | Most of my child's needs were met | 4 (44.4%) |
| | Only few of my child's needs were met | 3 (33.3%) |
| | None of my child's needs were met | 0 (0.0%) |
| | N | 9 |
| | Missing | 3 |
| Willingness to | No, definitely not | 1 (11.1%) |
| recommend the syrup to<br>another parent | Not really | 1 (11.1%) |
| | Yes, generally | 2 (22.2%) |
| | Yes, definitely | 5 (55.6%) |
| | N | 9 |
| | Missing | 3 |
| Satisfaction with<br>nformation received from | Quite dissatisfied | 0 (0.0%) |
| the IFU to use this<br>treatment | Indifferent or mildly dissatisfied | 0 (0.0%) |
| | Mostly satisfied | 6 (66.7%) |
| | Very satisfied | 3 (33.3%) |
| | N | 9 |
| | Missing | 3 |
| Ease of use of the syrup | No, definitely not | 0 (0.0%) |
| Lase of use of the syrup | Not really | 0 (0.0%) |
| | Yes, generally | 2 (22.2%) |
| | Yes, definitely | 7 (77.8%) |

| C1735 | Statist | tical Analysis Report | 14/05/2025 | Page <b>74</b> on <b>81</b> |
|---|---|---|---|---|
| | _ | | | |
| | | N | | 9 |
| | | Missing | | 3 |
| Feeling that the | | No, definitely not | | 0 (0.0%) |
| enjoyed the tas<br>syrup | ite of the | Not really | | 0 (0.0%) |
| | | Yes, generally | | 2 (22.2%) |
| | | Yes, definitely | | 7 (77.8%) |

<sup>\*3</sup> patients did not complete the satisfaction questionnaire (patients prematurely discontinued from the study)

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>75</b> on <b>81</b> |
|---|---|---|---|

Listing 17: Parents' satisfaction (D3 or D4) (FAS population) (n=12 with 3 missing satisfaction questionnaires)

| Listing 17: Pa | rents | satistaction | Listing 17: Parents satisfaction (D3 or D4) (FAS population) (n=12 with 3 missing satisfaction questionnaires) | population) ( | 7 = 1 | ر<br>الالا | missing sausiacile | on questioninaire | (S) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient<br>number | FAS | SAFETY | PERFORMANCE | Inclusion<br>Date | Age | Sex | Questionnaire<br>date | Day of completion | ۵ | 02 | ဗ | Φ | Q5 | 90 |
| 6D9E.102 | Yes | Yes | Yes | 14/03/2024 | 5.3 | Girl | 17/03/2024 | Day 4 | Good | Most of my<br>child's needs<br>were met | Yes,<br>definitely | Mostly<br>satisfied | Yes,<br>definitely | Yes,<br>definitely |
| 6D9E.109 | Yes | Yes | No | 25/03/2024 | 1.5 | Girl | | | | | • | | | • |
| 6D9E.111 | Yes | Yes | No | 28/03/2024 | 2.3 | Girl | 31/03/2024 | Day 4 | Poor | Only few of my<br>child's needs<br>were met | No,<br>definitely<br>not | Mostly<br>satisfied | Yes,<br>generally | Yes,<br>generally |
| 6D9E.112 | Yes | Yes | Yes | 28/03/2024 | 3 | Boy | | | | | | | | |
| 6D9E.113 | Yes | Yes | Yes | 28/03/2024 | 4.3 | Воу | 31/03/2024 | Day 4 | Good | Most of my<br>child's needs<br>were met | Yes,<br>generally | Mostly<br>satisfied | Yes,<br>definitely | Yes,<br>definitely |
| 6D9E.114 | Yes | Yes | Yes | 29/03/2024 | 3.9 | Girl | 01/04/2024 | Day 4 | Excellent | Almost all of my child's needs were met | Yes,<br>definitely | Mostly<br>satisfied | Yes,<br>definitely | Yes,<br>definitely |
| 6D9E.116 | Yes | Yes | Yes | 03/04/2024 | 0.7 | Boy | 06/04/2024 | Day 4 | Excellent | Almost all of my child's needs were met | Yes,<br>definitely | Very<br>satisfied | Yes,<br>definitely | Yes,<br>definitely |
| 6D9E.118 | Yes | Yes | Yes | 04/04/2024 | 9 | Girl | 07/04/2024 | Day 4 | Good | Most of my<br>child's needs<br>were met | Yes,<br>definitely | Mostly<br>satisfied | Yes,<br>definitely | Yes,<br>definitely |
| 6D9E.127 | Yes | Yes | ON | 02/10/2024 | 5.6 | Girl | 05/10/2024 | Day 4 | Good | Only few of my<br>child's needs<br>were met | Yes,<br>generally | Very<br>satisfied | Yes,<br>definitely | Yes,<br>definitely |
| 6D9E.129 | Yes | Yes | Yes | 14/10/2024 | 2.2 | Воу | 16/10/2024 | Day 3 | Good | Most of my<br>child's needs<br>were met | Yes,<br>definitely | Mostly<br>satisfied | Yes,<br>generally | Yes,<br>definitely |
| 6D9E.133 | Yes | Yes | No | 04/11/2024 | 0.7 | Воу | 07/11/2024 | Day 4 | Fair | Only few of my<br>child's needs<br>were met | Not<br>really | Very<br>satisfied | Yes,<br>definitely | Yes,<br>generally |
| 6D9E.134 | Yes | Yes | No | 06/11/2024 | 2.1 | Girl | | | | | | | | |

Q1. Quality of therapeutic management received by the child Q2. Response to the child's needs Q3. Willingness to recommend the syrup to another parent Q4. Satisfaction with information received from the IFU to use this treatment Q5. Ease of use of the syrup Q6. Feeling that the child enjoyed the taste of the syrup

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>76</b> on <b>81</b> |
|---|---|---|---|
|---|---|---|---|

### 4.13 Secondary outcome: Safety evaluation - SAFETY population

Table 13 : Adverse events – Summary of AEs (SAFETY)

| | All patie | ents (SAFETY) |
|---|---|---|
| Safety | | N=12 |
| | # events | # patients (%) |
| Number of patients with at least one: | | |
| Adverse events (AEs) | 7 | 4 (33.3%) |
| Serious Adverse Events (SAEs) | 0 | 0 (0.0%) |
| Adverse Device Effect (ADE): related to procedures | 2 | 1 (8.3%) |
| Adverse Device Effect (ADE): related to device | 2 | 1 (8.3%) |
| Serious Adverse Device Effect (SADE): related to procedures | 0 | 0 (0.0%) |
| Serious Adverse Device Effect (SADE): related to device | 0 | 0 (0.0%) |
| AEs leading to dose or frequency modifications | 0 | 0 (0.0%) |
| AEs leading to temporary treatment discontinuation | 0 | 0 (0.0%) |
| AEs leading to permanent treatment discontinuation | 1 | 1 (8.3%) |
| AEs leading to the need of concomitant treatment | 4 | 2 (16.7%) |
| SAEs leading to permanent treatment discontinuation | 0 | 0 (0.0%) |
| SAEs leading to the need of concomitant treatment | 0 | 0 (0.0%) |
| Non-serious AEs | 7 | 4 (33.3%) |
| AEs leading to death | 0 | 0 (0.0%) |
| SAE leading to death | 0 | 0 (0.0%) |
| Treatment-related AEs leading to death | 0 | 0 (0.0%) |
| | 0 | 8 (66.7%) |
| | 1 | 1 (8.3%) |
| | 2 | 3 (25%) |
| | 3 | 0 (0.0%) |
| | 4-8 | 0 (0.0%) |
| | >8 | 0 (0.0%) |
| Number of adverse events (AE) per patient | N | 12 |
| | Missing | 0 |
| | Mean (± SD) | $0.6 \pm 0.9$ |
| | Median | 0 |
| | Q1-Q3 | 0 - 1.5 |
| | Min – Max | 0 - 2 |
| | 0 | 11 (91.7%) |
| | 1 | 0 (0.0%) |
| Number of ADE per patient: related to procedure | 2 | 1 (8.3%) |
| | 3 | 0 (0.0%) |
| | 4-8 | 0 (0.0%) |

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>77</b> on <b>81</b> |
|---|---|---|---|
| | | >8 | 0 (0.0%) |
| | | N | 12 |
| | | Missing | 0 |
| | | Mean (± SD) | $0.2 \pm 0.6$ |
| | | Median | 0 |
| | | Q1-Q3 | 0 - 0 |
| | | Min – Max | 0 - 2 |
| | | 0 | 11 (91.7%) |
| | | 1 | 0 (0.0%) |
| | | 2 | 1 (8.3%) |
| | | 3 | 0 (0.0%) |
| | | 4-8 | 0 (0.0%) |
| Normala | on of ADE non-mations, related to device | >8 | 0 (0.0%) |
| Numb | er of ADE per patient: related to device | N | 12 |
| | | Missing | 0 |
| | | Mean (± SD) | $0.2 \pm 0.6$ |
| | | Median | 0 |
| | | Q1-Q3 | 0 - 0 |
| | | Min – Max | 0 - 2 |

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>78</b> on <b>81</b> |
|---|---|---|---|

| $\overline{}$ |
|---------------|
| ິທ |
| ≐ |
| $\Box$ |
| Φ |
| = |
| $\sigma$ |
| Q |
| 4 |
| 4 |
| Įo. |
| 0 |
| 4 |
| Ä |
| = |
| ч |
| _ |
| ٠ |
| Ш |
| ۳ |
| ĄE |
| z |
| Ч |
| = |
| ਛ |
| ō |
| sting |
| ₩ |
| S |
| 1 <u>8</u> .F |
| ÷: |
| ω |
| $\Box$ |
| $\simeq$ |
| .= |
| isting |
| .22 |
| _ |

| | ( d | | | |
|---|---|---|---|---|
| Subject ID | 6D9E.111 | 6D9E.127 | 6D9E.133 | 6D9E.134 |
| Presence of the patient in the FAS population | Yes | Yes | Yes | Yes |
| Presence of the patient in the SAFETY population | Yes | Yes | Yes | Yes |
| Presence of the patient in the PERFORMANCE population | No | No | No | No |
| Date of inclusion | 28/03/2024 | 02/10/2024 | 04/11/2024 | 06/11/2024 |
| Age calculated in years | 2.3 | 5.6 | 0.7 | 2.1 |
| Sex (D1) | Girl | Girl | Boy | Girl |
| Number of adverse events per child | 2 | 2 | 2 | 1 |
| El 1 : 1st adverse event | VOMITING | HEAVY FATIGUE | DOSAGE ERROR | TONSILLITIS |
| MedDRA Primary System<br>Organ Class Term text for the<br>1st adverse event | GASTROINTESTINAL<br>DISORDERS | GENERAL DISORDERS AND<br>ADMINISTRATION SITE<br>CONDITIONS | INJURY, POISONING AND PROCEDURAL COMPLICATIONS | RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS |
| MedDRA Preferred Term text for the 1st adverse event | VOMITING | FATIGUE | UNDERDOSE | TONSILLITIS |
| Onset date for the 1st adverse event | 30/03/2024 | 03/10/2024 | 06/11/2024 | 07/11/2024 |
| End date for the 1st adverse event | 31/03/2024 | 05/10/2024 | 06/11/2024 | 07/11/2024 |
| AE duration, AE for the 1st adverse event | 1 | 2 | 0 | 0 |
| Intensity for the 1st adverse event | Moderate | · | | Moderate |
| El 2 : 2nd adverse event | INCREASED COUGH | INTENSE SORE THROAT | PRODUCT UNDERDOSING DUE<br>TO INCORRECT PIPETTE<br>HANDLING | |
| MedDRA Primary System<br>Organ Class Term text for 2nd<br>adverse event | RESPIRATORY, THORACIC AND<br>MEDIASTINAL DISORDERS | RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS | INJURY, POISONING AND PROCEDURAL COMPLICATIONS | |
| MedDRA Preferred Term text for 2nd adverse event | соисн | OROPHARYNGEAL PAIN | DEVICE USE ERROR | |
| Onset date for 2nd adverse event | 30/03/2024 | 03/10/2024 | 06/11/2024 | |
| End date for 2nd adverse event | 31/03/2024 | 05/10/2024 | 06/11/2024 | |
| AE duration, AE # for 2nd adverse event | 1 | 2 | 0 | |

### C1735\_RAS\_1.0\_RNSR\_20250514.docx

| _ |
|-----------------------------|
| Page <b>79</b> on <b>81</b> |
| 14/05/2025 |
| Statistical Analysis Report |
| C1735 |

| Statistical Analysis Report | 14/05/2025 | Page <b>80</b> on <b>81</b> |
|-----------------------------|------------|-----------------------------|
|-----------------------------|------------|-----------------------------|

### 4.14 Secondary outcome: Device deficiencies (SAFETY)

Table 14 : Device deficiencies - SAFETY population

| D | | All patients (SAFETY) |
|---|---|---|
| Device deficiencies | | N=12* |
| | N | 9 |
| <b>-</b> | Missing | 3 |
| The bottle damaged during the use | No | 9 (100.0%) |
| | Yes | 0 (0.0%) |
| _ | N | 9 |
| The plants decreased decises the con- | Missing | 3 |
| The pipette damaged during the use | No | 9 (100.0%) |
| | Yes | 0 (0.0%) |
| _ | N | 9 |
| Jse of more or less than the prescribed dose due to | Missing | 3 |
| difficulty using the pipette | No | 8 (88.9%) |
| | Yes | 1 (11.1%)** |
| _ | N | 9 |
| Jse of more or less than the prescribed dose due to | Missing | 3 |
| Use of more or less than the prescribed dose due to lack of clarity in the IFU | No | 9 (100.0%) |
| | Yes | 0 (0.0%) |
| _ | N | 9 |
| Eye and/or ear damage during use | Missing | 3 |
| | No | 9 (100.0%) |
| | Yes | 0 (0.0%) |
| | N | 9 |
| Child potentially allergic to syrup | Missing | 3 |
| | No | 9 (100.0%) |
| | Yes | 0 (0.0%) |
| _ | N | 9 |
| Someone else, other than the child used the syrup | Missing | 3 |
| Someone else, other than the child used the syrup (including accidental use) | No | 9 (100.0%) |
| | Yes | 0 (0.0%) |
| _ | N | 9 |
| Child accidently accesses the bottle | Missing | 3 |
| Clinic accidently accesses the dottle | No | 9 (100.0%) |
| | Yes | 0 (0.0%) |
| _ | N | 9 |
| Other pipette used than the one proposed | Missing | 3 |
| | No | 9 (100.0%) |

| C1735 | Statistical Analysis Report | 14/05/2025 | Page <b>81</b> on <b>81</b> |
|---|---|---|---|
|---|---|---|---|

| Davies deficiencies | All patients (SAFETY) | |
|--------------------------|-----------------------|------------|
| Device deficiencies | | N=12* |
| | Yes | 0 (0.0%) |
| | N | 9 |
| Syrup reached air tube | Missing | 3 |
| | No | 9 (100.0%) |
| | Yes | 0 (0.0%) |
| | N | 9 |
| Pipette reached air tube | Missing | 3 |
| | No | 9 (100.0%) |
| | Yes | 0 (0.0%) |

<sup>\*3</sup> patients did not complete the device deficiencies questionnaire (patients prematurely discontinued from the study)

\*\* patient 133 with misuse (cf AE section)